CLINICAL TRIAL: NCT05589259
Title: A Novel Treatment Approach to Complex Regional Pain Syndrome (CRPS): A Feasibility Study of Combined Peripheral Nerve Block and Physiotherapy
Brief Title: Feasibility Study of Combined Peripheral Nerve Block and Physiotherapy for CRPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tracy Cupido (Other)
Responsible Party: Sponsor-Investigator, Tracy Cupido, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRPS-BP-PT
Record Dates: First submitted 2022-09-24; First posted 2022-10-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Complex Regional Pain Syndromes
Keywords: chronic pain; pain management
MeSH Terms: conditions — Complex Regional Pain Syndromes; Chronic Pain; Agnosia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Axillary Brachial Plexus Block plus Physiotherapy (Experimental): Participants who are randomized to the experimental group (EXP arm) will receive a single-shot axillary-approach brachial plexus block with 1.5mg/kg (up to 50mg total) bupivacaine 0.25% at the Kingston Health Sciences Centre Chronic Pain Clinic (KHSC-CPC). Prior to treatment, a blinded third party will perform a baseline physical exam. Under the brachial plexus block, the physiotherapist will provide standard of care, including manual therapy. The patient will then complete a 6-week physiotherapy program, including GMI. Following the 6 week program, a blind observer will repeat the physical exam.
  Interventions: Procedure: Axillary Brachial Plexus Block plus Physiotherapy
- Physiotherapy alone (Active Comparator): Participants who are randomized to not receive a block (CON arm) will also have a baseline physical exam performed by a blinded third party. Following baseline data collection, the physiotherapist will provide standard of care, including manual therapy. They will then complete a 6-week home exercise program, including GMI. Following the 6 week program, a blinded observer will repeat the physical exam.
  Interventions: Procedure: Physiotherapy alone

INTERVENTIONS:
Procedure: Axillary Brachial Plexus Block plus Physiotherapy — Participants will receive a single-shot axillary-approach brachial plexus block. For the procedure, a 22g or larger peripheral intravenous cannula will be placed, and skin will be sterilized with chlorhexidine. Using aseptic technique, the anesthesiologist will anesthetize the skin and tract with 5cc of 1% lidocaine using a 25g 1.5" needle. After this, a 50mm 21g Pajunk needle will be guided under ultrasound with an in-plane technique to anesthetize the median, ulnar, radial, and musculocutaneous nerves. Identification of the axillary artery, vein and surrounding vessels will be done to ensure an intravascular injection is avoided. Once proper location is confirmed, the anesthesiologist will aspirate to ensure the needle is not intravascular. Once aspiration is confirmed negative, bupivacaine 0.25% 1.5mg/kg (lean body weight) will be injected in divided doses.
  30 minutes after placement of the block, the standardized physiotherapy protocol will begin.
  Arms: Axillary Brachial Plexus Block plus Physiotherapy
Procedure: Physiotherapy alone — Participants in the EXP arm and the CON arm will complete the same physiotherapy program.
  PHYSIOTHERAPY PROTOCOL The physiotherapy program will include manipulation with or without a block. The goal of manipulation is to break up adhesions, possibly overcoming microvascular dysfunction. After the manipulation, participants will take part in a 6-week program which will include a weekly one-hour session with a physiotherapist at the KHSC-CPC and a home exercise program (HEP). During each session, the physiotherapist will work with the participants to increase ROM and limb function using manual therapy, stretching, and strengthening exercises specific to the affected joint(s) and most importantly using GMI. At the end of each session, the physiotherapist will prescribe exercises to complete at home.
  Arms: Physiotherapy alone

SUMMARY:
Chronic pain is a debilitating condition affecting 1 in 5 Canadians with a yearly economic cost of over $40 billion in healthcare spending and loss of productivity. Since the prevalence of chronic pain is increasing, especially as the population ages, effective low-cost treatment is key to reduce the impact of chronic pain on patient quality of life and on healthcare costs. Due to the complexity of chronic pain and differences between the multitudes of pain conditions, developing effective treatments is challenging. This is especially true for Complex Regional Pain Syndrome (CRPS).

CRPS is characterized by severe pain out of proportion to tissue trauma, with local autonomic and inflammatory changes. The severity of pain from CRPS may result in an inability to work, depression, sleep disorders, or suicidal ideation.

Although its prevalence is low in Canada, CRPS is considered one the most debilitating and least understood pain conditions. As most current treatment options have low evidence of effectiveness, there is no definitive treatment available and most often, patients are struggling to maintain an acceptable quality of life. Thus, there is a pressing need to identify new and improved treatments for adults with CRPS.

An early hypothesis of CRPS pathophysiology posited that sympathetic nervous system over-activity led to many of the signs and symptoms of CRPS. As such, sympathetic nerve blocks, including stellate ganglion and lumbar sympathetic blocks, have been repeatedly investigated as a potential treatment of CRPS. However, a recent meta-analysis suggests that these blocks provided no benefits for those suffering with CRPS. Newer evidence suggests that a peripheral microvascular dysfunction may underlie CRPS pathophysiology. However, no clinical trials have investigated the efficacy of a treatment targeting this peripheral pathway.

The goal of this project is to assess the efficacy of a single-shot axillary approach to the brachial plexus block plus physiotherapy as a novel treatment protocol for CRPS. Our primary hypothesis is that providing a brachial plexus block in conjunction with a physiotherapy program would be superior to physiotherapy alone in treating pain and function in CRPS. Since this is a novel treatment protocol for CRPS, the purpose of our proposed study is to determine the feasibility of conducting a fully powered clinical trial.

DETAILED DESCRIPTION:
Chronic pain is a debilitating condition affecting 1 in 5 Canadians with a yearly economic cost of over $40 billion in healthcare spending and loss of productivity. Since the prevalence of chronic pain is increasing, especially as the population ages, effective low-cost treatment is key to reduce the impact of chronic pain on patient quality of life and on healthcare costs. Due to the complexity of chronic pain and differences between the multitudes of pain conditions, developing effective treatments is challenging. This is especially true for Complex Regional Pain Syndrome (CRPS).

CRPS is characterized by severe pain out of proportion to tissue trauma, with local autonomic and inflammatory changes. The severity of pain from CRPS may result in an inability to work, depression, sleep disorders, or suicidal ideation.

Although its prevalence is low in Canada, CRPS is considered one the most debilitating and least understood pain conditions. As most current treatment options have low evidence of effectiveness, there is no definitive treatment available and most often, patients are struggling to maintain an acceptable quality of life. Thus, there is a pressing need to identify new and improved treatments for adults with CRPS.

An early hypothesis of CRPS pathophysiology posited that sympathetic nervous system over-activity led to many of the signs and symptoms of CRPS. As such, sympathetic nerve blocks, including stellate ganglion and lumbar sympathetic blocks, have been repeatedly investigated as a potential treatment of CRPS. However, a recent meta-analysis suggests that these blocks provided no benefits for those suffering with CRPS. Newer evidence suggests that a peripheral microvascular dysfunction may underlie CRPS pathophysiology. However, no clinical trials have investigated the efficacy of a treatment targeting this peripheral pathway. Current evidence of the efficacy of peripheral nerve block in treating CRPS are mostly derived from small case studies involving cost- and labour-intense regimens, including in-patient protocols with continuous nerve blocks.

The goal of this project is to assess the efficacy of a single-shot axillary brachial plexus block plus physiotherapy as a novel treatment protocol for CRPS. Our primary hypothesis is that providing a brachial plexus block in conjunction with a physiotherapy program would be superior to physiotherapy alone in treating pain and function in CRPS. Since this is a novel treatment protocol for CRPS, the purpose of our proposed study is to determine the feasibility of conducting a fully powered clinical trial. The specific aims of the feasibility trial are to assess: 1) the capacity (recruitment and staffing) required for conducting a fully powered trial, 2) the design of the novel treatment protocol, and 3) the patient response to treatment and trial protocol.

Statement of Relevance The incidence of CRPS in the US is estimated to be 5.4-26.2 per 100,000 person-years. Although unknown, the incidence of CRPS in Ontario is likely similar considering similar prevalence of chronic pain with the US. CRPS is known to be severely debilitating, leading to decreased quality of life and substantial lost productivity, which can be long-term if not quickly and properly treated. Historically, proposed treatments have been variable, resource intensive and results have been mixed. Therefore, specialized pain clinics in Ontario and across Canada are struggling to provide effective and quality care for this patient population. To date there is no definitive treatment for CRPS. Thus, pain specialists have no other choice to trial several treatment options to possibly find one beneficial for their patients.

By testing the efficacy of a single shot brachial plexus block followed by physiotherapy, on an outpatient basis, with the combination of home-based structured physiotherapy, the investigators hope to define a reproducible and effective outpatient treatment for CRPS. If the investigators can demonstrate superiority of a brachial plexus block with physiotherapy over physiotherapy alone, the investigators will be laying the groundwork for further research into not only a new treatment protocol of CRPS that is feasible and scalable for pain clinics in Ontario and around the world but also translating animal models of CRPS pathophysiology to humans.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Meets the Budapest criteria for CRPS of the upper extremity
* Able to consent to treatment.

Exclusion Criteria:

* Allergy to local anesthetic
* Allergy to chlorhexidine
* Infection at site of injection
* Previous treatment of current CRPS with a regional anesthetic technique within 6 months
* Unable to tolerate regional anesthesia or physiotherapy
* Another pain condition that affects the same limb
* Patient refusal or inability to consent.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Assessment | 2 years
  Assess the ability to recruit 60 patients (30 per arm) to complete the study protocol.
  Protocol data: Attrition (with reasons) will be monitored by the research coordinator. Data completeness will be computed from data entered from surveys and electronic diaries. Treatment compliance data (visit attendance and average hours/day of home exercise completed weekly) will be collected.
  Staff time will be monitored using logs by each team member (e.g., physician, physiotherapist, blind assessor, nurses).
  Patient satisfaction: A custom patient satisfaction questionnaire will also be completed with post-treatment clinical assessment questionnaire to capture patients' impression of the study protocol (e.g., time commitment, treatment length).

SECONDARY OUTCOMES:
Cost | 2 years
  Estimate the cost of a randomized controlled study in order to apply for future funding.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No